CLINICAL TRIAL: NCT05070208
Title: Multicenter Retrospective Observatory of Patients With Acute Myeloid Leukemia to Core Binding Factor
Acronym: RETRO-CBF
Status: Completed | Type: Observational
Sponsor: Acute Leukemia French Association (Other)
Responsible Party: Sponsor
Other Study IDs: RETRO-CBF
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloblastic Leukemia Core Binding Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: NOT PROVIDED — NOT PROVIDED

SUMMARY:
Acute Core Binding Factor leukemias represent a specific category of acute myeloid leukemias that share prognostic factors, a specific mutational profile, and a favorable response to chemotherapy. Their management now follows the reference pattern from the French trial CBF-2006 closed to inclusions since November 2010. This includes intensive chemotherapy and intensification by allogeneic marrow transplant depending on the residual disease measured by RT qPCR . These leukemias have not been the subject of multicenter clinical trials since that date.

The results of this treatment regimen need to be evaluated. Known prognostic factors such as signaling mutations, clonal interference or residual disease follow-up (MRD) will be analyzed and updated in this recent cohort. The interaction between residual disease and mutational profile will be evaluated on the prognosis. Treatment with gemtuzumab-ozogamycin and first-line allogeneic transplantation will be investigated, depending on prognostic factors including associated mutations and residual disease. The course and early treatment of molecular relapses will be analyzed. The treatment and prognosis of cytological relapses will be described with in particular the role of tyrosine kinase inhibitors and therapeutic intensification.

DETAILED DESCRIPTION:
NOT PROVIDED

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosis of acute myeloid leukemia with CBF confirmed by cytogenetics (karyotype and / or FISH): t (8; 21), inv (16) or t (16; 16) and / or molecular biology (RUNX1-RUNX1T1 fusions or CBFB-MYH11)
* Initial management by intensive chemotherapy, hypomethylants or targeted therapies

Exclusion Criteria:

- Opposition expressed to research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Core Binding Factor Acute Myeloid Leukemia
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | December 2010 to December 2020

SECONDARY OUTCOMES:
- Complete remission rate (CR / CRp) | December 2010 to December 2020
- Overall survival (OS), relapse free survival (DFS) +/- censored with allogeneic transplant | December 2010 to December 2020
- Cumulative incidence of relapse (CIR) +/- censored at allograft | December 2010 to December 2020
- Second complete remission rate, OS, EFS, DFS and CIR post-relapse | December 2010 to December 2020
-Prognostic impact on OS, CR, EFS, DFS and CIR of recurrent somatic mutations | December 2010 to December 2020
- Interaction between mutations and MRD on OS, CR, EFS, DFS and CIR | December 2010 to December 2020
- Cumulative incidence of molecular relapse. | December 2010 to December 2020
- Prognostic impact on OS, CR, EFS, DFS, CIR and post-relapse survival of using first-line GO and relapsing | December 2010 to December 2020

CONTACTS AND LOCATIONS:
Overall Officials: ITZYKSON Raphael, Dr, Principal Investigator — SAINT LOUIS PARIS
Locations (26):
- France (26):
  - Chu Amiens, Amiens
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - AP-HP-GHU - Hôpital AVICENNE, Bobigny
  - CHU de la cote de Nacre, Caen
  - CH Métropole Savoie, Chambéry
  - Hôpital MILITAIRE PERCY, Clamart
  - Centre hospitalier Sud Francilien, Corbeil-Essonnes
  - Henri Mondor Aphp, Créteil
  - Dijon Chu, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay
  - LENS CHR, Lens
  - CHU, Lille
  - Limoges Chu, Limoges
  - CHU La Conception, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU Nice,Hopital Archet 1, Nice
  - Hopital Pitié-Salpétrière APHP, Paris
  - Hôpital Necker - APHP, Paris
  - Hôpital Saint Louis- APHP, Paris
  - Saint Antoine, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier de Roubaix, Roubaix
  - Centre Hospitalier de St Quentin, Saint-Quentin
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No